CLINICAL TRIAL: NCT06046677
Title: Investigation Into the Transcriptomic and Functional Profile of SEPsis in ONCology Patients
Brief Title: Sepsis in Oncology Patients
Acronym: SEPONC
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5669
Record Dates: First submitted 2023-06-08; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sepsis in Cancer Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat & PMBCs PAXgene RNA Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis cohort: Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.
  Organ dysfunction can be identified as an acute change in total SOFA score ≥2 points consequent to the infection.
  Interventions: Other: No intervention
- Elective cohort: Elective pre-operative upper GI surgical patients or elective stem cell transplant patients will be consented and enrolled at baseline, immediately prior to these procedures. If they go on to develop sepsis within 60 days of their surgery, they will go on to be sampled as per the sepsis cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The overall objective of this prospective observational study is to address the significant knowledge gap that exists around the impact of immune dysfunction on the development and survival from sepsis in patients with cancer. This proposal primarily focuses on establishing the transcriptomic immune profiles of sepsis patients with a background of cancer. This analysis will be complemented with in vitro functional analyses, and in addition will commence a collection of genome-wide data, including a focus on predicting white cell number and function in health. Uniquely, the investigators propose to establish a robust link between these analyses: transcriptomic, in vitro, and genome-wide, to enable them to comprehensively explore septic oncology patient 'immune phenotypes' and effectively identify novel exploitable therapeutic pathways.

To this end, this project will collect, analyse and/or sequence DNA, RNA, leukocytes and soluble materials from a cohort of oncology patients presenting to intensive care with sepsis. This cohort will include all-comers with an oncological background but will also focus on two core groups at high risk of sepsis where baseline samples can also be sought prior to major immunosuppressive events in the cancer pathway. These are:

1. Oesophageal/upper gastrointestinal (GI) cancer patients prior to systemic anticancer therapy initiation or surgery
2. Haematological malignancy patients prior to stem cell transplantation.

These sub-cohorts will provide a previously unexplored unique insight into the role of pre-existing patient transcriptomic phenotypes.

DETAILED DESCRIPTION:
The specific aims will be to perform multi-modal parallel immune phenotyping to determine:

* The transcriptomic (RNA) phenotypes (or 'signatures') of cancer patients with sepsis
* The association of these transcriptomic phenotypes with:

  1. Leukocyte function in sepsis, as quantified by cell surface and functional assays and plasma soluble mediator content
  2. Pre-existing genomic determinants such as leukocyte numbers
  3. Severity of, and outcome from, sepsis in oncology patients

ELIGIBILITY:
Sepsis cohort: Inclusion Criteria:

* Patients admitted to ICU with a diagnosis of sepsis as per 'Sepsis-3' definitions with a SOFA score [REF] ≥2 secondary to infection from any source
* ≥18 years of age
* Written consent from patient, personal or professional consultee, or deferred consent if none of the above available at admission

Sepsis cohort Exclusion Criteria:

• Death deemed imminent by the clinical team

Elective cohort inclusion criteria

* Patients undergoing elective major upper GI surgery (oesophago+/-gastrectomy) or stem cell transplant for haematological malignancy
* ≥18 years of age
* Written consent from patient

Elective cohort exclusion criteria

• Limitations in place regarding provision of treatment and/or organ support e.g., palliative patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who develop sepsis on ICU or require admission to ICU with sepsis will be identified and screened for enrolment by the research team at the Royal Marsden NHS Foundation Trust
  Elective pre-operative upper GI surgical patients or elective stem cell transplant patients will be consented and enrolled at baseline, immediately prior to these procedures.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Identification of circulating leukocyte transcriptomic phenotypes relating to mortality in sepsis patients with a background of cancer, (in comparison to those previously identified in non-immunosuppressed patients). | end of trial (4 years)
  Identification of circulating leukocyte transcriptomic phenotypes relating to mortality in sepsis patients with a background of cancer, (in comparison to those previously identified in non-immunosuppressed patients).
28 day mortality | end of recruitment (3 years)
  28 day mortality

SECONDARY OUTCOMES:
Differences in the trajectory of transcriptomic phenotypes of patients admitted to ICU with sepsis, and how they relate to severity scorings and mortality/morbidity outcomes | end of trial (4 years)
  how they relate to severity scorings and mortality/morbidity outcomes
Differences in the trajectory of functional phenotypes of patients admitted to ICU with sepsis, and how they relate to severity scorings and mortality/morbidity outcomes | end of trial (4 years)
  how they relate to severity scorings and mortality/morbidity outcomes
Differences in the trajectory of genomic phenotypes of patients admitted to ICU with sepsis, and how they relate to severity scorings and mortality/morbidity outcomes | end of trial (4 years)
  how they relate to severity scorings and mortality/morbidity outcomes
Identification of differences in transcriptomic phenotypes between patient subgroups and on comparison to non-immunosuppressed sepsis patients. Comparison in length of stay measures and quality of life parameters | end of trial (4 years)
  Comparison in length of stay measures and quality of life parameters
Identification of differences in functional phenotypes between patient subgroups and on comparison to non-immunosuppressed sepsis patients. Comparison in length of stay measures and quality of life parameters | end of trial (4 years)
  Comparison in length of stay measures and quality of life parameters
Identification of differences in genomic phenotypes between patient subgroups and on comparison to non-immunosuppressed sepsis patients. Comparison in length of stay measures and quality of life parameters | end of trial (4 years)
  Comparison in length of stay measures and quality of life parameters

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No